CLINICAL TRIAL: NCT03707704
Title: Quality Control of an In-hospital Strengthening Protocol in Spinal Cord Injured Subjects During Initial Rehabilitation - a Prospective Observational Study
Brief Title: Quality Control of a Strengthening Protocol in Subjects With Spinal Cord Injury
Acronym: MKraft_Erstr
Status: Completed | Type: Observational
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Other Study IDs: 2018-16
Record Dates: First submitted 2018-10-11; First posted 2018-10-16 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Spinal Cord Injury, Acute
Keywords: Exercise; Rehabilitation
MeSH Terms: conditions — Spinal Cord Injuries; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SCI patients in primary rehabilitation

SUMMARY:
The aim of the master's thesis is to evaluate the clinic-internal strengthening concept of the Swiss Paraplegic Centre (SPZ). The SPZ is a rehabilitation clinic for spinal cord injured people. The strengthening concept has been routinely used since 2015.

By default, the patients complete - depending on which training phase they are in - three to four strength training sessions per week. As part of the master's thesis, the development of maximum strength of patients with spinal cord injury (SCI) in primary rehabilitation will be studied. It is explicitly taken care of that the patients comply with the training requirements. Furthermore, factors which prevent a consistent buildup of strength - such as medical complications (pressure sores, pneumonia, urinary tract infections) - are systematically recorded.

The findings should provide information on the effect and qualitative transfer of the existing strength concept in everyday clinical practice. The strength training performed is accompanied by the master student and documented in a standardized manner.

ELIGIBILITY:
Inclusion Criteria:

* Patients in initial rehabilitation
* SCI Level C1-C5 (ASIA Score C-D)
* SCI Lever C6-L5 (ASIA Score A-D)
* Traumatic and non-traumatic SCI
* Disease-related paraplegia, high-grade stenoses and central cord Syndromes
* Age >= 18 years
* The maximum force is tested on three predefined training devices, two devices for the upper and a device for the lower extremity. The participants will only be included in the study if they are capable of succeeding in at least both exercises for the upper extremity

Exclusion criteria:

* Polyneuropathic diseases such as Critical Illness and Guillain Barré Syndrome
* Degenerative diseases such as multiple sclerosis and amyotrophic lateral sclerosis etc.
* Cognitive impairments
* Compliance of less than 2/3 of the training sessions
* ≥ 14 days without training
* more than 6 weeks between assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with acute spinal cord injury during their initial rehabilitation
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
One-repetition-maximum as parameter for the maximum force [kg] | Change from 0 weeks to 5 weeks and from 5 weeks to 10 weeks
  Calculated one-repetition-maximum based on the Brzycki equation formula

SECONDARY OUTCOMES:
Number of completed training sessions (training compliance) | Change from 0 weeks to 5 weeks and from 5 weeks to 10 weeks
  Number of completed training sessions per participant
Causes of study exclusion | From 0 weeks to 10 weeks
  Systematic documentation of exclusion causes during the participation in the study

CONTACTS AND LOCATIONS:
Locations (1):
- Swiss Paraplegic Centre, Nottwil, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No